CLINICAL TRIAL: NCT03340987
Title: Clinical Evaluation of the Amount of Root Coverage Following The Use of VISTA Technique Versus Coronally Advanced Flap in Combination With Subepithelial Connective Tissue Graft for Management of Multiple Gingival Recessions: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of the Amount of Root Coverage Following The Use of VISTA Technique Versus Coronally Advanced Flap in Combination With Subepithelial Connective Tissue Graft for Management of Multiple Gingival Recessions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Walaa Shaaban, B.Sc. in Oral and Dental Medicine, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: VISTA technique RCT
Record Dates: First submitted 2017-09-21; First posted 2017-11-14 (Actual); Last update posted 2018-07-06 (Actual); Status verified 2018-07

CONDITIONS: Gingival Recession
Keywords: vestibular incision subperiosteal tunnel access; coronally advanced flap; subepithelial connective tissue graft; multiple gingival recessions
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vista technique with SCTG (Experimental): vestibular incision subperiosteal tunnel access combined with subepithelial connective tissue graft
  Interventions: Procedure: vestibular incision subperiosteal tunnel access
- coronally advanced flap with SCTG (Active Comparator): coronally advanced flap combined with subepithelial connective tissue graft
  Interventions: Procedure: Coronally advanced flap

INTERVENTIONS:
Procedure: vestibular incision subperiosteal tunnel access — vertical vestibular incision will be made down to the periosteum followed by creating a tunnel without reflecting the interdental papilla. Then a free gingival graft will be optained from the palate and de-epithelialized extraorally. The connective tissue graft will then be applied through the tunnel and the gingival margin will be sutured and the sutures will be fixed to the tooth surface by flowable composite. Then the vestibular incision will be sutured.
  Other Names: Vista technique
  Arms: Vista technique with SCTG
Procedure: Coronally advanced flap — Two horizontal incisions will be made mesial and distal to the recession area followed by two oblique incisions extended to the alveolar mucosa and a full-split thickness flap will be elevated. De-epithelialization will be done to receive the connective tissue graft obtained from the palate by de-epithelializing a free gingival graft. Then the flap will be advanced coronally aand sutured without tension
  Other Names: CAF
  Arms: coronally advanced flap with SCTG

SUMMARY:
Patients with multiple recession defects will be randomly oriented into to groups. The test group will recieve a relatively new technique, the VISTA technique, combined with connective tissue graft that will be harvested from the palate. The control group will recieve coronally advanced flap with connective tissue graft. subjects will be followed up for 6 months after the surgery. Any complications, that may occur, will be dealt with.

DETAILED DESCRIPTION:
The aim of the study is to evaluate the effectiveness of the VISTA technique with subepithelial connective tissue graft for management of multiple gingival recessions compared to the coronally advanced flap with subepithelial connective tissue graft.

• Research hypothesis: Null hypothesis: There is no difference in the amount of root coveragefollowing VISTA technique when comparingVISTA technique versus coronally advanced flap combined with subepithelial connective tissue graft.

Trial design:

* Blinded, Randomized controlled trial
* 2 arms:

  1. Intervention:

     VISTA technique with connective tissue graft
  2. Control:

     Coronally advanced flap with connective tissue graft.

     Study setting:
     * Study is to be conducted in theOralMedicine and Periodontology department,Faculty of Oraland Dental Medicine - Cairo University, Egypt.
     * Patients are to be selected from the outpatient clinic of the department of OralMedicine and Periodontology-Cairo University.

     Clinical Examination Clinical periodontal parameters included; recession depth, recession width, width of keratinized gingiva, gingival thickness, plaque index, gingival index, probing pocket depth and clinical attachment loss. These parameters will be recorded using Williams graduated periodontal probe at three sites for all teeth, mesiobuccal, midbuccal and distobuccal (except for recession width) to nearest millimeters. Measurements will be reported at base line and at 3 & 6 months postoperatively months).

     Radiographic Examination:

     Intraoral periapical radiographs will be taken at the time of the initial examination to confirm the diagnosis of Miller's class I or II.

     Clinical photographs:

     Clinical photographs will be taken at baseline, during surgery and at 3 & 6 month postoperatively.

     Treatment protocol

     Pre-surgical phase:
     * Full mouth supragingival scaling and subgingival debridement will be performed using ultrasonic device and manual scalers and curettes.
     * Detailed instructions in self-performed plaque control measures will be given and the patients will be educated that maintenance of proper plaque control is of utmost concern.
     * The patients will be reevaluated four weeks after initial therapy to ensure their competence with the study design and recording the previously mentioned measurements.

     Surgical phase:

     A. Recipient site preparation with VISTA technique (Test group) • The VISTA approach as described by Zahdeh, 2011 begins with a vestibular access incision after administration of local anesthesia¹. The location of the access incision depends on the sites being treated.
     * The incision will be made through the periosteum to elevate a subperiosteal tunnel, exposing the facial osseous plate.
     * ¹ Artinisba 40 mg/0.01 mg/ml. Articaine (D.C.I) 40.00 mg hydrochloride, Epinephrine (D.C.I) (tartrate) 0.01 mg. Insibia Dental S.L.U.
     * This tunnel will extend at least one tooth beyond the teeth requiring root coverage to mobilize gingival margins and facilitate coronal repositioning. A periosteal elevator will be used to create the subperiosteal tunnel and introduced through the vestibular access incision and inserted between the periosteum and bone to elevate the periosteum, creating the subperiosteal tunnel.

     It is important to extend the tunnel elevation sufficiently beyond the mucogingival margin as well as through the gingival sulci of the teeth being augmented to allow for low-tension coronal repositioning of the gingiva.

     • Additionally, the subperiosteal tunnel will be extended interproximally under each papilla as far as the embrasure space permits, without making any surface incisions through the papillae.

     • After harvesting the subepithelial connective tissue graft, it will be carefully repositioned through the vestibular incision and well adapted below the gingival margin of each tooth.

     • The graft and mucogingival complex will then be advanced coronally and stabilized in the new position with a coronally anchored suturing technique. This technique entails placing a horizontal mattress suture using a 6.0 suture at approximately 2 to 3 mm apical to the gingival margin of each tooth.

     • If keratinized gingiva is present, the suture will be placed within the band of keratinized gingiva. The suture will be tied so that the knot is positioned at the midcoronal point of each tooth.

     • For wide teeth or when coronal repositioning creates excessive tension, an additional suture will be placed. Each tooth will then be prepared for attachment of the suture to the tooth.
     * The facial enamel surface of each tooth will be briefly etched for less than 5 seconds with acid etch, thoroughly washed, and dried. The gingival margin will be advanced coronally to the most coronal level of the interproximal papillae. If during coronal repositioning excessive tension is detected, the subperiosteal tunnel will be further elevated in all directions to facilitate mobilization of the marginal gingiva.
     * The sutures will be secured to the facial aspect of each tooth by placing a small amount of flowable composite resin over the knot, effectively preventing apical relapse of the gingival margin during the initial stages of healing.
     * The vestibular incision will then be approximated and sutured primarily with multiple interrupted sutures.
     * Sutures at the access incision will be removed after 1 week.
     * Coronally anchored bonded sutures will be removed 3-weeks postoperatively to allow for immobilization of the gingival margin during the initial phases of healing.

     B. Recipient site preparation with coronally advanced flap (CAF):

     In the control group, a CAF will be performed while preparing the recipient site according to de Sanctis and Zucchelli (2007) as follows; • Two horizontal incisions will be performed, mesial and distal to the recession defect located at a distance from the tip of the anatomical papillae equal to the depth of the recession plus 1-2 mm will be done. This will be followed by two beveled oblique, slightly divergent, incisions starting at the end of the two horizontal incisions and extending to the alveolar mucosa.

     • The resulting trapezoidal-shaped flap will be elevated with a full-split thickness approach.

     • Flap elevation will continue and scoring of all muscle attachments will be performed until it will be possible to move the flap passively in the coronal direction.

     • This will be done keeping the blade parallel to the external mucosal surface. The flap should be stable in its final coronal position even without the sutures.

     • The root surface will be mechanically treated with the use of periodontal curettes. It must be considered that only the portion of the root exposure with loss of clinical attachment will be instrumented.
     * The facial soft tissue of the anatomic interdental papillae coronal to the horizontal incisions will be de-epithelized to create connective tissue beds upon which the coronally advanced flap will be sutured.

     C. Harvesting subepithelial connective tissue graft:

     A subepithelial connective tissue graft (SCTG) will be harvested from the palate using Zucchilli's technique (zucchelli, 2010):

     • A free epithelialized gingival graft will be obtained. This will be done by performing two horizontal incisions; the coronal one is 1-1.5 mm away from the gingival margin.
     * Along the coronal horizontal incision, the blade will be held perpendicular to the bone and once the adequate soft tissue thickness is obtained, the blade is oriented parallel to the superficial surface to separate the free gingival graft.
     * The thickness of the graft will be maintained uniform while proceeding apically with the blade.
     * Once the graft is separated, any fatty tissues will be removed.
     * The graft will then be de-epithelialized extra orally.

     Postoperative Care:

     Postoperative medication
* Administration of:

  1. Postoperativeoral analgesic (Brufen® 400 mg t.d.s) ² will be prescribed to the patients for the first 3 days then whenever needed. Systemic antibiotic will be prescribed (Amoxicillin® 500mg t.d.s) ³ for one week to prevent postsurgical infection.

  2. Patients will be instructed to rinse with Hexitol® oral rinse ⁴ twice daily for 2 weeks.(Dandu & Murthy, 2016).

  ² Ibuprofen 600 mg, Kahira Pharm. & Chem. Ind. Co. Egypt, Underlicence from: Abbott Laboratories

  ³ Amoxicillin 500mg Misr Co. for pharmaceutical industries, for: OCTOBER PHARMA S.A.E. - EGYPT.

  ⁴Hexitol, CHLORHEXIDINE HCL 0.125%.THE ARAB DRUG COMPANY (ADCO) - A.R.E
* Patient self-care instructions:

  3. Subjects will be instructed to avoid excessive muscle tractioning or trauma to the treated areas for the first 3 weeks and told not to brush teeth involved in the surgery.

After 3 weeks the resorbable sutures will be removed. Three weeks post surgically the patients will be instructed to gently brush the operated area with a soft tooth brush using roll technique.

Follow-up and Criteria of Evaluation:

Clinical Evaluation:

Each patient will be evaluated at 1, 3, and 6 months post-operatively (Lafzi et al, 2016).

Criteria for Discontinuing or Modifying Intervention:

Intervention will be discontinued or modified according to events.

Strategies to improve adherence to intervention:

Patients will be recalled every 3 months for supportive periodontal therapy.

Concomitant care:

The patients will receive postoperative instructions and oral hygiene guidelines that should be followed during the follow-up period.

Sample size Sample size was calculated in the Evidence-based Dentistry Center, Faculty of Oral and Dental Medicine, Cairo University.

A total sample size of 26 (13 per group) including drop outs.

Recruitment strategy:

* Patients will be selected from the outpatient clinic of the Oral Medicine and Periodontology Department, Faculty of Oraland Dental Medicine-Cairo University
* Screening of patients will continue until the target sample is achieved.
* Identifying and recruiting potential subjects will be achieved through patient database.

Allocation

Allocation: random sequence generation:

Methods of generating randomization:

Patients will be randomly selected using computer generated randomization (www.randomizer.org) and will be performed by another individual other than the investigator. The numbers will be allocated to each patient.

Allocation - concealment mechanism The two groups will be equally prepared for surgical implant placement. Then the decision of whether immediate implant with simultaneous soft tissue grafting or immediate implant placement onlywill be made according to the randomized numbers in a sequentially numbered, opaque, sealed envelope. The number will be picked by the supervisor.

Implementation

* All patients who provide an informed consent for participation as well as fulfill the inclusion criteria will be randomized.
* The supervisor will generate the allocation sequence as well as assign the participants to the intervention. The investigator will enroll the participants.

Blinding Due to the nature of the procedures, it's not possible to blind the principal investigator for neither the treatment protocol nor the participant. The outcome evaluators and data analysts will be blinded to group assignment. Detailed instructions on methods to maintain the blinding procedure will be given to the researchers and outcome evaluators.

Data collection, management and analysis

Data collection method:

The phone numbers and address of the patient included in the study will be recorded from them or extracted from the patient's file.

Plans to promote participant retention and complete follow- up

* Telephone numbers of all patients included the study will be recorded as a part of the written consent.
* All patients will be given a phone call at the time of the pre-determined follow up dates.

Data management

* All data will be entered and saved electronically.
* Patient files are to be stored in numerical order and stored in secured file. Data will be encrypted using a password.
* All data will be maintained after completion of the study.

Statistical method

Statistical methods for analyzing primary, secondary and tertiary outcomes:

Data will be analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 21 (SPSS Inc. Chicago, IL). Numerical data will be described as mean and standard deviation or median and range or interquartile range, as appropriate. Categorical data will be described as numbers and percentages. The data will be explored for normality using Kolmogrov-Smirov test and Shapiro-Wilk test. Comparisons between two groups and over time will be done by 2 way analysis of variance for repeated measures.

If the time factor is not considerable, comparisons between the two groups for normally distributed numeric variables will be done using the Student's t-test while for non-normally distributed numeric variables will be done by Mann-Whitney test.

A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two tailed.

ELIGIBILITY:
Inclusion Criteria:

* Patient with two or more adjacent teeth with Miller class I or II facial gingival recessions.
* Good oral hygiene
* Accepts follow-up period (cooperative patients).
* Patient provides a signed informed consent.

Exclusion Criteria:

* Patients with systemic disease that may affect periodontal health and healing.
* Current and former smokers
* Pregnant females.
* Subjects received any surgical periodontal therapy in the area of interest for minimum of 6 months prior to the study.
* Subjects taking drugs known to interfere with wound healing.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Estimated)
Dates: Start 2018-08 (Estimated); Primary Completion 2019-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Amount of root coverage | 6 months
  complete root coverage after surgical correction measured in millimeters by using periodontal probe

SECONDARY OUTCOMES:
Root Coverage Esthetic score a numbering score | 6 months
  a system to evaluate esthetics after surgical root coverage giving a numbering score by a periodontal probe
Clinical Attachment level gain in millimeters | 6 months
  the clinical attachment level is the measurement of the position of the soft tissue in relation to the cemento-enamel junction (CEJ) that is a fixed point that does not change throughout life. Two measurements are used to calculate the CAL: the probing depth and the distance from the gingival margin to the CEJ. measured using a periodontal probe in millimeters.
Width of Keratinized tissue in millimeters | 6 months
  It is measured from the mucogingival junction (MGJ) to the free gingival margin. The MGJ will be identified using the roll technique. Measured in millimeters using a periodontal probe
Probing depth in millimeters | 6 months
  It is measuring the distance from the base of pocket to the gingival margin. The probe will be inserted parallel to the long axis of the tooth using light force. Measured in millimeters using a periodontal probe
Gingival thickness in millimeters | 6 months
  It will be measured by penetrating the gingiva mid-buccally in the attached gingiva, half way between mucogingival junction and free gingival groove (Goaslind et al. 1977) with the periodontal probe after giving local anesthesia to measure the thickness of gingival tissues. Measured in millimeters using a periodontal probe
Post-Operative Pain a numerical rating scale | 2 weeks
  Numerical Rating Scale (NRS) with numbers from 0 to 10 ('no pain' to 'worstpain imaginable')for the first 2 weeks postoperatively.
Post-Operative Swelling verbal rating scale | 7 days
  Verbal Rating Scale (VRS); absent(no swelling), slight (intraoral swelling at the operated area), moderate (moderate intraoral swelling at the operated area) and intense (intensive extraoral swelling extending beyond the operated area), assessed during the first 7 postoperative days
Post-Surgical Patient Satisfaction numerical rating scale | 6 months
  A numerical rating scale will be used. A 3-item questionnaire is asked and the patients shall use a 7 point answer scale.

IPD SHARING:
Plan to Share IPD: Undecided